CLINICAL TRIAL: NCT04810767
Title: Prevalence and Risk Factors for Chronic Pain After Cesarean Delivery in Upper Egypt: Retrospective Study
Brief Title: Chronic Pain After CS in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bahaa Mohammed Refaie (Other)
Responsible Party: Sponsor-Investigator, Bahaa Mohammed Refaie, Lecturer of anesthesia and ICU, Sohag University
Organization: Sohag University (Other)
Other Study IDs: 2020
Record Dates: First submitted 2021-03-21; First posted 2021-03-23 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Pain experienced assessed by questionnaire described by Nikolajsen et al, 2004

SUMMARY:
This retrospective study will include Women who will attending to Azhar assuit, Sohag and South valley universities hospitals for any reason in the duration from 1 May to 31 October 2021, and who underwent elective CD under spinal anesthesia with horizontal lower abdominal surgical incision within last two years.

Exclusion criteria will be refusal to participate, age less than 18 years, recent CD (within 3 months), if the infant had died, and history of chronic pain medications or psychiatric disorder.

Data collection

Participants will be contacted personally by one of study authors. Data collected are consisted of:

* Participants' characteristics as Age, parity and ways of delivery, weight, height, residency, husband smoking status, work, previous abdominal surgery, history of diabetes mellitus and hypertension.
* Last CD related data which include presence of multiple pregnancies, if CD was in private/public facility, presence surgical wound infection.
* Pain experienced will be assessed by questionnaire described by Nikolajsen et al, 2004

ELIGIBILITY:
Inclusion Criteria:

* Women attending to Azhar assuit, Sohag and South valley universities hospitals for any reason in the duration from 1 May to 31 October 2021, and who underwent elective ceserean section under spinal anesthesia with horizontal lower abdominal surgical incision within last two years

Exclusion Criteria:

* refusal to participate, age less than 18 years, recent ceserean section (within 3 months), if the infant had died, and history of chronic pain medications or psychiatric disorder

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 20-40 years old Women attending to Al Azhar assuit, Sohag and South valley universities hospitals for any reason in the duration from 1 May to 31 October 2021, and who underwent elective ceserean section under spinal anesthesia with horizontal lower abdominal surgical incision within last two years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Chronic pain | Three months after the last ceserean section
  Pain experienced assessed by questionnaire described by Nikolajsen et al, 2004

CONTACTS AND LOCATIONS:
Overall Officials: Kareem ElGebaly, Lecturer, Study Chair — Lecturer of anesthesia and ICU; Hossam Eldin Mostafa, Consultant, Study Director — Consultant of anesthesia and ICU Elhelal insurance hospital